CLINICAL TRIAL: NCT01073319
Title: Rivastigmine as a Treatment for Methamphetamine Dependence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Richard De La Garza, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: H-23064; R01DA023964 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2010-02-19; First posted 2010-02-23 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Methamphetamine Dependence; Substance Abuse; Methamphetamine Abuse
Keywords: Methamphetamine; Rivastigmine
MeSH Terms: conditions — Substance-Related Disorders | interventions — Sugars; Rivastigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Matching oral placebo capsule as control.
  Interventions: Other: Placebo
- Rivastigmine 3 mg (Active Comparator)
  Interventions: Drug: Rivastigmine
- Rivastigmine 6 mg (Active Comparator)
  Interventions: Drug: Rivastigmine

INTERVENTIONS:
Other: Placebo — Administration of placebo pill
  Other Names: Sugar pill
  Arms: Placebo
Drug: Rivastigmine — Participants will be randomized to rivastigmine (1.5 mg bid) for 6 days of each phase.
  Other Names: Exelon
  Arms: Rivastigmine 3 mg
Drug: Rivastigmine — Participants will be randomized to rivastigmine (3 mg bid) for 6 days of each phase.
  Other Names: Exelon
  Arms: Rivastigmine 6 mg

SUMMARY:
To study the effects of treatment with rivastigmine on craving produced by experimental administration of methamphetamine.

DETAILED DESCRIPTION:
We recently completed a double-blind placebo-controlled human laboratory study demonstrating that treatment with a low dose of the acetylcholinesterase (AChE) inhibitor rivastigmine reduced methamphetamine (METH)-induced craving (see Preliminary Studies, Fig. 2). This finding is consistent with the preclinical report indicating that the AChE inhibitor donepezil reduced METH-seeking behavior in rats following exposure to a non-contingent dose of METH (Hiranita et al. 2006). To extend our clinical findings, we propose a 3-year human laboratory study to evaluate effects of higher doses of rivastigmine on METH-induced craving and on self-administration of METH. Our recently completed work indicates that 3mg rivastigmine attenuated METH-induced craving in the laboratory. Given that higher dosages of this produce greater inhibition of nicotinic acetylcholine (ACh) receptors (in the treatment of Alzheimer's disease), it is reasonable to predict that 6mg and 12mg will have more pronounced effects on craving and other measures of reinforcement. This human laboratory study is a critical next step in the evaluation of rivastigmine as a potential treatment for METH dependence. We propose to include only participants exhibiting METH-induced craving by screening potential participants prior to admission (criterion based upon Preliminary Studies, Fig. 5). Selection of participants demonstrating METH-induced craving will facilitate assessment of effects of rivastigmine on craving. The project has the following objectives:

Primary Objective: To characterize the effects of treatment with rivastigmine (0, 3, and 6 mg) on craving produced by experimental administration of METH (0, 15 and 30mg, IV).

Secondary Objective: To characterize the effects of treatment with rivastigmine (0, 3, and 6 mg) on choices for METH exhibited in a self-administration paradigm (0 and 5mg, IV).

ELIGIBILITY:
Inclusion Criteria - In order to participate in the study, participants must:

* Be English-speaking volunteers who are not seeking abstinence-focused treatment at the time of the study
* Be between 18-55 years of age
* Meet DSM-IV-TR criteria for METH dependence
* Self-report that preferred route of METH use is intravenous or smoke
* Have vital signs as follows: resting pulse between 50 and 90 bpm, blood pressures between 85-150 mmHg systolic and 45-90 mmHg diastolic
* Have a breathalyzer test indicating an undetectable blood alcohol level upon admission
* Have hematology and chemistry laboratory tests that are within normal ("b10%) limits with the following exceptions: a) liver function tests (total bilirubin, ALT, AST, and alkaline phosphatase) < 3 x the upper limit of normal, and b) kidney function tests (creatinine and BUN) < 2 x the upper limit of normal
* Have a baseline ECG that demonstrates normal sinus rhythm, normal conduction, and no clinically significant arrhythmias
* Have a medical history and brief physical examination demonstrating no clinically significant contraindications for study participation, in the judgment of the admitting physician/ Nurse Practitioner (or Advanced Practice Nurse) and the PI
* Weigh between 60 and 100 kg
* Have a negative urine drug screen, with the exception of methamphetamine or marijuana

Exclusion Criteria - Potential participants will be excluded from participation in the study if any of the following apply:

* Have any previous medically adverse reaction to METH, including loss of consciousness, chest pain, or epileptic seizure
* Have neurological or psychiatric disorders, as assessed by MINI, such as: a. episode of major depression within the past 2 years; b. lifetime history of schizophrenia, other psychotic illness, or bipolar illness; c. current organic brain disease or dementia assessed by clinical interview; d. history of or any current psychiatric disorder which would require ongoing treatment or which would make study compliance difficult; e. history of suicide attempts within the past three months and/or current suicidal ideation/plan; and f. history of psychosis occurring in the absence of current METH use
* Meet DSM-IV criteria for dependence on alcohol or other drugs, except for nicotine or marijuana
* Have evidence of clinically significant heart disease or hypertension as determined by the admitting physician/NP/APN
* Have evidence of untreated or unstable medical illness including: neuroendocrine, autoimmune, renal, hepatic, or active infectious disease
* Have HIV and are currently symptomatic, have a diagnosis of AIDS, or are receiving antiretroviral medication
* Be pregnant or nursing. Other females must either be unable to conceive (i.e., surgically sterilized, sterile, or post-menopausal) or be using a reliable form of contraception (e.g., abstinence, birth control pills, intrauterine device, condoms, or spermicide). All females must provide negative pregnancy urine tests before study entry, and weekly throughout the study
* Have any history of asthma, chronic coughing and wheezing, or other chronic respiratory illnesses
* Currently use alpha or beta agonists, theophylline, or other sympathomimetics
* Have any other illness, condition, or use of medications, which in the opinion of the PI and/or the admitting physician/NP/APN would preclude safe and/or successful completion of study.

Criteria for Discontinuation Following Initiation:

Participants will be discharged if they have a positive breath test indicating use of alcohol or a urine test indicating illicit use of drugs while in the GCRC, if they do not comply with study procedures, or if they do not tolerate METH. All female subjects of child bearing potential will be tested for pregnancy at each admission and those with positive test results will be discharged.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Effects of rivastigmine and methamphetamine on cardiovascular measures
  Beginning with intake, vital signs (temperature with orthostatic BP and HR) will be recorded every 8 hours. Before and after the intravenous METH infusion, subjects' physiologic responses will be closely monitored using repeated HR, BP, and ECG readings.

SECONDARY OUTCOMES:
Effects of rivastigmine and methamphetamine on subjective measures (craving and choices for METH)
  Effects of treatment with rivastigmine on craving produced by experimental administration of METH (0, 15 and 30mg, IV) will be measured using a computerized visual analogue scale (VAS), designed to provide rapidly acquired ratings of METH-induced craving, dysphoria, and euphoria. VAS measures will be collected prior to METH administration and at 5, 10, 15, 20, 30, 45, 60, 90, and 120 min following METH administration. Effects of treatment with rivastigmine on choices for METH (0 and 5mg) will be assessed using an existing model of drug self-administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States